CLINICAL TRIAL: NCT01286935
Title: A Phase III, Double-blind, Placebo-controlled, 18-mon Ext Study Long-term Efficacy & Safety of 50 & 100mg/Day Doses of Safinamide, as add-on Therapy, in Idiopathic PD Pts With Motor Fluctuations, Treated With Levodopa, Who May be Receiving DA, and/or Anticholinergic
Brief Title: 18-month Study of Long-term Efficacy & Safety of Safinamide as add-on Therapy in Patients With Mid-late Stage PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Dr Ravi Anand (Chief Medical Officer), Newron Pharmaceuticals S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-1015/018/III/2006; 2006-005861-21 (EudraCT Number)
Record Dates: First submitted 2010-08-23; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; PD; Levodopa; Patients with idiopathic Parkinson's Disease with motor fluctuations,
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (50mg/day) (Experimental)
  Interventions: Drug: Safinamide
- High Dose (100mg/day) (Experimental)
  Interventions: Drug: Safinamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Safinamide
  Arms: Low Dose (50mg/day)
Drug: Safinamide
  Arms: High Dose (100mg/day)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the long-term efficacy and safety of two doses of safinamide (50 and 100 mg/day, p.o), compared to placebo, as add-on therapy in patients with idiopathic Parkinson's disease with motor fluctuations, who are currently receiving a stable dose of levodopa.

ELIGIBILITY:
Inclusion Criteria:

* The patient completed 24 weeks of treatment in Study 016, or, if the patient discontinued prematurely, he/she returned for scheduled efficacy evaluations at Weeks 12 and 24, as part of the Retrieved Dropout (RDO) population.
* The patient was compliant with taking study medication in Study 016.
* The patient is willing to participate in the study and signed an approved Informed Consent form.

Exclusion Criteria:

* The patient is experiencing clinically significant adverse events that would put the patient at risk for participating in the study.
* The patient has shown clinically significant deterioration during participation in Study 016, and has reached Hoehn and Yahr Stage V.
* The patient discontinued Study 016 prematurely for any reason, and did not return for scheduled efficacy evaluations at Weeks 12 and 24.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Mean change in the dyskinesias rating scale (DRS) during "on" time | Up to 104 weeks (from baseline 016 to EOS study 018)
  mean change in the dyskinesias rating scale (DRS) during "on" time from baseline (study 016) to endpoint (last visit in study 018).

SECONDARY OUTCOMES:
Endpoints include 'ON time', responder rates and UPDRS IV change | Up to 104 weeks (from baseline 016 to EOS study 018)
  * Chge in ON time (ON+ON minor dysk),
  * Diary Resp Rate at 12-m, 18 & 24 m on the ITT&mITT pop&pts who completed 2-yr period
  * UPDRS IV chge in total score,items 32-35 & 32-34
  * Time develop tblsome dysk(> 30min incr of tblsome dysk)
  * Time develop any (minor &/or tblsome) dysk (> 30 min incr of dysk)
  * Chge ADLs during ON, vs pbo(UPDRS II)
  * Maintenance of effect in UPDRS II "resp'(resp >=20% impr in ADLs).
    * chge in L-dopa dose
    * chge in any PD(other than L-dopa)drug dose
  * Chge in UPDRS III, CGI-C and CGI-S
  * Chge in diary categories(ON, OFF, ON minor dysk, ON tblsome dysk, ASLEEP)

CONTACTS AND LOCATIONS:
Overall Officials: See Study 016 for details, Principal Investigator — PI's are the same as for study NW-1015/016/III/2006

REFERENCES:
- See also: Related Info — http://www.newron.com/